CLINICAL TRIAL: NCT03737357
Title: A Randomized Controlled Study to Assess Intra-patient Clinical Performance of Dental Implants With a SLActive® vs. SLA® Surface
Brief Title: Dental Implants With a SLActive® vs. SLA® Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR 2017-05
Record Dates: First submitted 2018-10-25; First posted 2018-11-09 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-02

CONDITIONS: Partially Edentulous Patients
Keywords: dental implants; SLActive® surface; biomarkers; BLT implant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLActive® implant (Experimental)
  Interventions: Device: SLActive® implant
- SLA® implant (Active Comparator)
  Interventions: Device: SLA® implant

INTERVENTIONS:
Device: SLActive® implant — One study test (SLActive® surface) (and simultaneously, in a split-mouth design one study control (SLA® surface) implant (Bone Level Tapered, Roxolid®)) will be placed in two different quadrants of partially edentulous patients. The implants will be placed at premolars, molars and canine positions in the mandible and maxilla (healed extraction sites). Implants will be restored with a single crown or splinted restorations 8 weeks after implant placement.
  Arms: SLActive® implant
Device: SLA® implant — One study test (SLActive® surface) (and simultaneously, in a split-mouth design one study control (SLA® surface) implant (Bone Level Tapered, Roxolid®)) will be placed in two different quadrants of partially edentulous patients. The implants will be placed at premolars, molars and canine positions in the mandible and maxilla (healed extraction sites). Implants will be restored with a single crown or splinted restorations 8 weeks after implant placement.
  Arms: SLA® implant

SUMMARY:
This post-market study is to show that dental implants with a SLActive® surface (SLActive® implants) show non-inferior clinical performance compared to dental implants with a SLA® surface (SLA® implants). The primary hypothesis is that 12 months after implant loading, the bone loss around the SLActive® implants will not be appreciably greater than around the SLA® implants.

The occurrence of adverse events and device deficiencies will also be recorded to confirm once more the safety of the Straumann® Bone Level Tapered (BLT), Roxolid® implant.

Osseointegration and anti-inflammatory potential of SLActive® implants will be evaluated in the study as secondary endpoints.

DETAILED DESCRIPTION:
This is a prospective, single-blinded, randomized, paired sample, multi-center clinical study. Eight visits per patient are scheduled in this study. The final analysis will be conducted after all patients completed the 12-month visit.

The study devices are CE- (Conformité Européenne, meaning European Conformity) marked products and used within their intended use.

Two centers in Spain will participate.

ELIGIBILITY:
Inclusion Criteria:

* males and females, at least 18 years old
* partially edentulous patients in need of two or more dental implants (canine to molars) placed in two different quadrants in healed sites (3 months post extraction)
* subject must have voluntarily signed the informed consent, is willing and able to attend scheduled follow-up visits, and agrees that the encoded data will be collected and analyzed

Exclusion Criteria:

* any contraindications for oral surgical procedures
* dental implant placement contraindicated according to Instructions for Use (IFU)
* subjects with inadequate oral hygiene (FMPS ≥ 20%)
* subjects who are currently heavy smokers (defined >10 cigarettes per day or >1 cigar per day) or who use chewing tobacco
* subjects with drug or alcohol abuse
* patients requiring soft tissue and bone grafting procedures
* inadequate bone volume
* severe bruxism or clenching habits
* women who are pregnant or planning to become pregnant at any point during the study duration.
* patients who have systemic factors that could interfere with the healing process of either bone or soft tissue or the osseointegration process (e.g. bone metabolism disturbances, uncontrolled diabetes mellitus, anticoagulation drugs/ hemorrhagic diatheses)
* patients with local factors that could interfere with the healing process, such as untreated periodontal diseases, acute infection of implant site, temporomandibular joint disorders, treatable pathologic diseases of the jaw and changes in the oral mucosa)
* conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, Prof. Dr., Principal Investigator — Professor and Chairman of Periodontology; Juan Blanco-Carrión, Prof. Dr., Principal Investigator — Professor in Periodontology
Locations (2):
- Spain (2):
  - Universidad Complutense, Madrid
  - Universidad de Santiago de Compostela, Santiago de Compostela

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened at 2 investigational centers in Spain
Pre-assignment Details: A total of 70 patients were screened. Of those, 68 subjects were enrolled
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | SLActive® Implant | SLA® Implant
Started | 68; 68 Implants | 68; 68 Implants
Completed | 61; 61 Implants | 61; 61 Implants
Not Completed | 7; 7 Implants | 7; 7 Implants

BASELINE CHARACTERISTICS:
Population: This study used a split-mouth design. Each participant received both SLActive® and SLA® implants. As a result, the same 68 participants appear under both arms. The Total column reflects the number of unique participants (N=68).
Units Other Than Participants: Implants
Groups:
- Total: Total of all reporting groups
Arm/Group | SLActive® Implant | SLA® Implant | Total
Number analyzed (Participants) | 68 | 68 | 68
Number analyzed (Implants) | 68 | 68 | 136
Age, Continuous [Median (Full Range); unit: years] | 56 [26 to 79] | 56 [26 to 79] | 56 [26 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 33 | 33 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian | 0 | 0 | 0
  Ethnicity: European | 67 | 67 | 134
  Ethnicity: Other | 1 | 1 | 2
Smoking status (never, past, current) [Count of Participants; unit: Participants]
  Never smoked | 26 | 26 | 52
  Past smoker (<10 years since cessation) | 13 | 13 | 26
  Past smoker (>=10 years since cessation) | 19 | 19 | 38
  Current smoker (<= 10 cigarettes per day) | 10 | 10 | 20
  Current smoker (1 cigar per day) | 0 | 0 | 0
  Current smoker (> 10 cigarettes per day) | 0 | 0 | 0
  Current smoker (>1 cigar per day) | 0 | 0 | 0
  Current smoker (e-cigs) | 0 | 0 | 0
Number of missing teeth [Mean (Standard Deviation); unit: Teeth] | 10.5 (4.9) | 10.5 (4.9) | 10.5 (4.9)
Number of Implants [Mean (Standard Deviation); unit: Implants] | 1.2 (1.9) | 1.2 (1.9) | 1.2 (1.9)
Number of planned implants [Mean (Standard Deviation); unit: Implants] | 3.1 (1.0) | 3.1 (1.0) | 3.1 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Bone Level Change 12 Months After Implant Loading
Description: The primary efficacy objective of this study was to confirm the performance of the SLActive® implants by means of bone level change 12 months after implant loading, as described in the CIP (CR2017-05, v03).
Time Frame: 12 months after implant loading
Population: Per protocol Population: defined as each eligible study subject with one study control and one study test implant and who performed all follow-up visits.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SLActive® Implant | SLA® Implant
Number analyzed (Participants) | 55 | 55
mm | 0.214 (0.391) | 0.056 (0.093)
Statistical Analysis 1: Comparison: SLActive® Implant vs SLA® Implant; Test type: Non-Inferiority — The tolerance range or non-inferiority margin characterizes the largest absolute difference which is considered to be dismissible. A MBL of less than 0.5mm within the first year after implant loading constitutes an acceptable clinical standard(10, 18, 19). In this clinical trial, a non-inferiority margin of 20% of the acceptable clinical standard was chosen, which amounts to 0.1mm; p = 0.074, t-test, 1 sided; Non-inferiority one-sided paired t-tests using a non-inferiority margin of -0.10mm; paired difference = 0.01 — The paired difference is (SLActive® bone level change from baseline (CFB) - SLA® CFB (i.e. resorption)); In the PP population, the paired difference between SLActive® and SLA® bone level change from baseline (CFB) was estimated at 0.01 mm with a standard deviation of 0.444 mm (95% CI: -Inf, 0.11; p = 0.074), based on a one-sided paired t-test with a non-inferiority margin of 0.10 mm

2. Primary Outcome: Occurrence of Adverse Device Effects and Device Deficiencies That Could Have Led to a Serious Adverse Device Effect
Description: Occurrence of adverse device effects and device deficiencies that could have led to a serious adverse device effect
Time Frame: 12 months after implant loading
Population: The SAF populations defined as all patients who were enrolled in the study and who received a study device
Measure: Number; unit: events
Arm/Group | SLActive® Implant | SLA® Implant
Number analyzed (Participants) | 68 | 68
events
  Number of ADE | 14 | 20
  Number of DD | 0 | 0

3. Secondary Outcome: Change in Inflammatory and Anti-inflammatory Biomarkers Concentrations
Description: Change in inflammatory and anti-inflammatory biomarkers (IL-10, IL-4, IL-6, IL-1beta, TNF-alpha, IL-2) concentrations in gingival crevicular fluid samples.
Time Frame: At implant placement, 1 and 4 weeks after implant placement
Population: Intention To Treat (ITT) population: each eligible and randomized study patient who received control and test implants in two different quadrants and from whom at least one follow-up measurement after placement is available.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | SLActive® Implant | SLA® Implant
Number analyzed (Participants) | 68 | 68
picograms per milliliter
  Inflammation (IL-6) at implant placement | 437.4 (1056.2) | 508.3 (1296.7)
  Inflammation (IL-6) at implant Week 4 | 17.2 (77.4) | 8.6 (38.5)
  Inflammation (IL-1B) at implant placement | 11.3 (26.8) | 8.4 (17.2)
  Inflammation (IL-1B) at Week 4 | 29.2 (65.8) | 35.2 (88.1)
  Inflammation (TNF-a) at implant placement | 13.3 (36.4) | 13.0 (30.1)
  Inflammation (TNF-a) at Week 4 | 14.2 (25.7) | 20.1 (46.3)
  Inflammation (IL-2) at implant placement | 1.9 (3.1) | 1.7 (2.8)
  Inflammation (IL-2) at Week 1 | 0.4 (0.5) | 0.9 (2.0)
  Anti-inflammation (IL-10) at implant placement | 18.3 (35.2) | 17.7 (44.4)
  Anti-inflammation (IL-10) at Week 4 | 22.5 (40.0) | 28.0 (51.3)
  Anti-inflammation (IL-4) at implant placement | 3.7 (7.3) | 5.7 (14.5)
  Anti-inflammation (IL-4) at Week 4 | 3.3 (3.6) | 3.6 (4.5)

4. Secondary Outcome: Change in Osseointegration Biomarkers Concentrations
Description: Change in osseointegration biomarkers ( VEGF, osteocalcin (OCN), osteopontin (OPN)) concentrations in gingival crevicular fluid samples.
Time Frame: 1, 2, 4 and 8 weeks after implant placement
Population: ITT population: each eligible and randomized study patient who received control and test implants in two different quadrants and from whom at least one follow-up measurement after placement is available.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | SLActive® Implant | SLA® Implant
Number analyzed (Participants) | 68 | 68
picograms per milliliter
  VEGF-a at implant placement | 39.3 (295.2) | 26.0 (272.7)
  VEGF-a at 4 weeks | 73.6 (504.4) | 28.6 (573.5)
  OCN at implant placement | 760.3 (1394.5) | 2408.6 (8935.4)
  OCN at 8 weeks | 159.8 (79.6) | 117.7 (76.3)
  OPN at implant placement | 6064.2 (11713.2) | 4419.0 (7887.0)
  OPN at 8 weeks | 939.3 (1677.1) | 876.6 (1789.8)

5. Secondary Outcome: Implant Survival
Description: Implant survival at 12 months after implant loading
Time Frame: 12 months after implant loading
Population: ITT population - defined as each eligible and randomized study patient who received control and test implants in two different quadrants and from whom at least one follow-up measurement after placement is available
Measure: Number; unit: number of lost implants
Arm/Group | SLActive® Implant | SLA® Implant
Number analyzed (Participants) | 68 | 68
number of lost implants | 3 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | SLActive® Implant | SLA® Implant
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 2/68 | 2/68
Other Adverse Events (participants affected / at risk) | 26/68 | 26/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SLActive® Implant (N=68) | SLA® Implant (N=68)
Anal fistula (Gastrointestinal disorders) | 1 | 1
Hernia (Nervous system disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLActive® Implant (N=68) | SLA® Implant (N=68)
Mechanical complications (Product Issues) | 6 (6) | 6 (6) — Including fracture/chipping of prosthesis; loosening of Abutment/Occlusal screw; Loss/failure of a healing cap; the crown doesn't fit
Biological Complications (General disorders) | 10 (10) | 10 (10) — Including bruising, local irritation and pain
Other complications (General disorders) | 3 (3) | 3 (3) — Including facial traumatism, loss of composite covering the crown, and transitory dizziness/nausea during procedure
Biological Complications - hard tissue related (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (9) — Including Early Loss/Failure Of Implant (I.E. Before Osseointegration); Implant Mobility (Tactile Horizontal Or Vertical; Late Loss/Failure Of Implant (I.E. After Osseointegration); Low Primary Stability (At Surgery)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT03737357/Prot_SAP_000.pdf